CLINICAL TRIAL: NCT03786692
Title: TH-138: Phase II Randomized Trial of Carboplatin + Pemetrexed + Bevacizumab, With or Without Atezolizumab in Stage IV Non-squamous NSCLC Patients Who Harbor a Sensitizing EGFR Mutation or Have Never Smoked
Brief Title: Phase II Randomized Trial of Carboplatin+Pemetrexed+Bevacizumab+/- Atezolizumab in Stage IV NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-138; 18-1077 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: The design of this study will be an open label, randomized, phase 2 study in adult (≥ 18 years) male and female subjects with stage IV disease who have never smoked, irrespective of their driver mutation status, as well as subjects who have tumors that possess a driver mutation.
  The study will be comparing the four agent treatment group (Arm A) that includes carboplatin + pemetrexed + bevacizumab + atezolizumab versus a three agent control group (Arm B) that includes carboplatin + pemetrexed + bevacizumab for 4 cycles, each cycle lasting for 3 weeks. Treatment will be followed by maintenance in both arms that will include all agents except carboplatin. There is no crossover in this study.
  1. Arm A: Carboplatin + Pemetrexed + Bevacizumab + Atezolizumab Maintenance: Pemetrexed + Bevacizumab + Atezolizumab
  2. Arm B: Carboplatin + Pemetrexed + Bevacizumab Maintenance: Pemetrexed + Bevacizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Arm A: Carboplatin + Pemetrexed + Bevacizumab + Atezolizumab Maintenance: Pemetrexed + Bevacizumab + Atezolizumab
  Interventions: Drug: Arm A
- Arm B (Active Comparator): Arm B: Carboplatin + Pemetrexed + Bevacizumab Maintenance: Pemetrexed + Bevacizumab
  Interventions: Drug: Arm B

INTERVENTIONS:
Drug: Arm A — Carboplatin + Pemetrexed + Bevacizumab + Atezolizumab
  Arms: Arm A
Drug: Arm B — Carboplatin + Pemetrexed + Bevacizumab
  Arms: Arm B

SUMMARY:
While cigarette smoking remains the primary cause of most lung cancer cases, lung carcinoma in never smokers account for nearly 20 percent of cases. Never smokers with lung cancer typically present with different molecular profiles from that of smokers, which results in prognostic and therapeutic implications. Molecular changes in NSCLC that have therapeutic significance include mutations in the epidermal growth factor receptor (EGFR) and rearrangements in the anaplastic lymphoma kinase (ALK) gene. These driver mutations typically are present in lung tumors found in never or light smokers.

The addition of bevacizumab to carboplatin and paclitaxel in first-line treatment of non-squamous NSCLC showed improved survival compared to carboplatin and paclitaxel alone, 12.3 vs. 10.3 months respectively. Results from the POINTBREAK trial demonstrated that carboplatin + pemetrexed + bevacizumab is an alternative option to carboplatin + paclitaxel + bevacizumab, with comparable survival but less toxicity. In recent years, immunotherapy has emerged as a form of treatment that can lead to robust responses in a subset of patients. The PD-1 inhibitor nivolumab and the PD-L1 inhibitor atezolizumab have shown prolonged survival in comparison to docetaxel in patients who previously progressed with chemotherapy, irrespective of PD-L1 expression. Thus, this study combines immunotherapeutic agent atezolozumab with an ant-angiogenic agent, bevacizumab, and double platinum therapy (carboplatin and pemetrexed).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed stage IV non-squamous non-small cell lung cancer
* Must have either tumors that harbor an EGFR mutation in exon 19 or exon 21, or must be never smoker wild-types. Never smoker wild-types are defined as patients with tumors without an ALK or ROS1 rearrangement, and are not harboring any EGFR mutation (this includes exons 19 or 21, exon 20, and any other rare EGFR mutations). Never smoker wild-type patients must have smoked less than 100 cigarettes in a lifetime. Patients with an EGFR mutation in exon 19 or 21 may be included irrespective of their smoking history. If a patient whose tumor originally had an exon 19 or 21 mutation develops a secondary activating or sensitizing mutation in exon 18-21 as a result of resistance to EGFR TKI therapy, then that patient is eligible. If tissue-based testing for EGFR mutation status is not available, blood-based EGFR testing that confirms presence of a mutation in exon 19 or 21 is acceptable, and these patients may be included in the stud
* Must have measurable disease by CT or MRI, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v 1.1
* Tumors that harbor an EGFR exon 19 or exon 21 mutation must have received prior treatments with one or more TKIs. A minimum washout period of 3 days is required to begin treatment in this trial. Patients who are never smoker wild-types must be treatment naïve
* Must be chemotherapy, anti-VEGF therapy alone, and immunotherapy naive, with the exception of prior oral TKIs which are required for EGFR mutated patients. Patients who have received prior anti-VEGF therapy in combination with a TKI for advanced stage EGFR-mutated disease may be included. The number of prior oral TKIs and duration of use is neither specified nor limited.
* History of treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  * No ongoing requirement for corticosteroids as therapy for CNS disease
  * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization
  * No clinical evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
  * New asymptomatic CNS metastases detected at the screening scan must be ≤1 cm in size with no prior radiation therapy. These patients may then be eligible without the need for an additional brain scan prior to randomization, if all other criteria are met
* May have received curative intent therapy (adjuvant therapy or therapy for locally advanced NSCLC), if this therapy was completed greater than 1 year from entry into the trial
* Age > 18 years
* ECOG performance status of 0 or 1
* Must have normal organ and marrow function as defined below. The use of G-CSF should follow standard recommendations and physician discretion. If blood transfusion is performed for achieving hemoglobin levels, the levels should stay at ≥ 9.0 mg/ml for at least a week after transfusion.

Absolute neutrophil count > 1,500/mcL Hemoglobin ≥ 9.0 mg/ml Platelets > 100,000/mcL Total bilirubin ≤1.5 X institutional upper limit of normal (ULN) AST/ALT (SGOT/SGPT) < 3 times institutional normal limits, or up to 5 times institutional normal limits if the patient has liver metastases Creatinine OR Creatinine clearance ≤1.5 X ULN, OR > 40 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal as per Cockcroft-Gault formula International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) <1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Thyroid stimulating hormone (TSH) Within normal limits a

a: If TSH is not within normal limits at baseline, the subject will still be eligible if total T3 or free T4 are within normal limits.

* Full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). If receiving warfarin, the patient must have an INR ≤3.0. For heparin and LMWH there should be no clinically significant active bleeding (with no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
* A biopsy, either core, cell block from FNA or cell block from surgical resection, must be available for the study. If the sample is not adequate, the patient must agree to provide a fresh biopsy specimen before the start of treatment. Any available archival tissue will also be collected. While a biopsy sample must be adequate and available for the study, an inadequate tissue sample would not be explicitly exclusionary and further discussion with the sponsor is allowed to assess the eligibility of the patient for the trial if, for clinical or other reasons, a new biopsy sample cannot be obtained.
* Urinary protein must be ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24 hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in the protocol).
* Females of child-bearing potential must be willing to use an effective method of contraception, for the course of the study through at least 6 months after the last dose of study medication.
* Males who have Women of Child-bearing Potential (WOCBP) partners must agree to use effective method of contraception for the course of the study through 8 months after the last dose of study medication.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Patients currently receiving any other investigational agents, immunomodulatory agents, chemotherapy, or TKIs. EGFR mutation-positive patients must have received prior TKI treatment
* Any Grade 3-4 GI bleeding within 3 months prior to first dose of protocol therapy.
* Untreated CNS metastases that are >1 cm in size are excluded, even if they are asymptomatic. Patients with treated brain metastases will be allowed if brain imaging obtained within 30 days of trial enrollment reveals stable disease.
* Cirrhosis at a level of Child-Pugh B or worse, or cirrhosis of any degree and a history of hepatic encephalopathy, or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
* Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol therapy.
* Uncontrolled or poorly-controlled hypertension (>150 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to randomization
* Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing wound, active ulcer, or untreated bone fracture within 28 days prior to first dose of protocol therapy
* Subjects with a history of smoking greater than a 100 cigarettes in a lifetime, unless their tumor has an EGFR exon 19 or exon 21 mutation.
* Patients with active, suspected, or known autoimmune disease that has required systemic treatment in the past one year (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Hormone replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patients with a history of hemoptysis (defined as bright red blood or ≥1/2 teaspoons) within 1 month prior to first dose of protocol therapy or with radiographic evidence of major blood vessel invasion or encasement by cancer.
* Undergone major surgery within 28 days prior to first dose of study treatment, or minor surgery/ subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
* Receiving chronic anti-platelet therapy other than aspirin, including non-steroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted. Occasional use of NSAIDs is allowed (for example daily use for less than a week; treating physician discretion is permitted to differentiate between occasional vs chronic use)
* Have not recovered from adverse events due to agents administered earlier except neuropathy and alopecia. Physician's discretion is allowed to decide which unresolved adverse events from previous therapy (for NSCLC) prohibit patient participation in this study.
* Requiring more than 10 mg prednisolone (or its equivalent) per day are excluded.
* Any evidence of interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or pneumonitis requiring oral or IV glucocorticoids. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with known latent or active tuberculosis infection are excluded.
* Have received a live vaccine within 30 days prior to cycle 1 Day 1.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (significant), cirrhosis, or psychiatric illness/ social situations that would limit compliance with the study requirements.
* Known history of testing positive for immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Known history of chronic hepatitis B virus infection or chronic hepatitis C virus indicating chronic infection that is not cured.
* Subjects with previous malignancies (except non-melanoma skin cancers, and in situ cancers, such as, bladder, gastric, colon, cervical/ dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study registration and no additional therapy is required or anticipated to be required during the study period.
* Leptomeningeal disease
* Uncontrolled tumor-related pain

  * Requiring pain medication must be on a stable regimen at study entry.
  * Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to randomization. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
  * Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for locoregional therapy, if appropriate, prior to randomization.
* Ca > 12 mg/dl or corrected serum calcium > ULN

  * Patients who are receiving denosumab prior to randomization must be willing and eligible to receive a bisphosphonate instead while in the study
* Pregnant or breast feeding
* Known hypersensitivity to Chinese hamster ovary cell products or any of the study drugs.
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Clear tumor infiltration into the thoracic great vessels is seen on imaging
* Clear cavitation of pulmonary lesions is seen on imaging
* Diagnosis of squamous cell carcinoma of the lung.
* Lung tumor with a known ALK or ROS1 rearrangement or an EGFR mutation other than in exon 19 or exon 21.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12.5 months
  Time a patient shows progression of disease from the time of intervention

SECONDARY OUTCOMES:
To perform a safety analysis in all treated subjects: NCI CTCAE v 5.0 | 15 months
  Observe safety of combination as per NCI CTCAE v 5.0
To compare the overall response rate (ORR) of Arm A to Arm B | 15 months
  ORR is defined as the portion of patients with partial or complete response as measured using RECIST 1.1 criteria
To compare the duration of response of Arm A to Arm B | 15 months
  Time from documentation of tumor response to disease progression, measured using RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bodor, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bodor JN, Patel JD, Wakelee HA, Levy BP, Borghaei H, Pellini B, Costello MR, Dowell JE, Finley G, Huang CH, Neal JW, Nieva JJ, Puri S, Socinski MA, Thomas C, Ross EA, Litwin S, Clapper ML, Treat J. Phase II Randomized Trial of Carboplatin, Pemetrexed, and Bevacizumab With and Without Atezolizumab in Stage IV Nonsquamous Non-Small-Cell Lung Cancer Patients Who Harbor a Sensitizing EGFR Mutation or Have Never Smoked. Clin Lung Cancer. 2023 Nov;24(7):e242-e246. doi: 10.1016/j.cllc.2023.05.003. Epub 2023 May 11. PMID 37451930